CLINICAL TRIAL: NCT06295549
Title: A Phase I, Open-label Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LUCAR-G39P, a Dual-targeted Cell Preparation Targeting CD19/CD20, in Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: Targeting CD19/CD20 Dual-targeted Cell in Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Achieve the proof of concept.
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2304-0001
Record Dates: First submitted 2024-02-18; First posted 2024-03-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2024-10

CONDITIONS: Relapsed and Refractory B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: LUCAR-G39P cells product (Experimental): Each subject will be given a single-dose LUCAR-G39P cells infusion at each dose level.
  Interventions: Biological: LUCAR-G39P cells product

INTERVENTIONS:
Biological: LUCAR-G39P cells product — LUCAR-G39P cells product Prior to infusion of the LUCAR-G39P, subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine

SUMMARY:
A phase I, open-label clinical study to evaluate the safety, tolerability, and efficacy of LUCAR-G39P, a dual-targeted cell preparation targeting CD19/CD20, in patients with relapsed/refractory B-cell non-Hodgkin lymphoma

DETAILED DESCRIPTION:
his is an open-label, dose-escalation/dose extension study to assess the safety, tolerability, and efficacy of LUCAR-G39P in the patient ≥ 18 years of age with relapsed or refractory B-cell non-Hodgkin lymphoma. Subjects who meet the eligibility criteria will receive a single dose of LUCAR-G39P injection. The study will include the following sequential phases: screening, pre-treatment (lymphodepleting chemotherapy), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have fully understood the possible risks and benefits of participating in this study, are willing to follow and able to complete all trial procedures, and have signed informed consent.
2. Aged 18-75 years (inclusive).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically confirmed B-cell non-Hodgkin Lymphoma that expresses at least one of CD19/CD20.
5. At least one evaluable tumor lesion according to Lugano 2014 criteria.

Response to prior therapy is consistent with one of the following:

1. Primary refractory.
2. Relapsed or refractory after 2 or more lines of therapy.
3. For LBCL, 3B FL. t-iNHL:

   * Relapse within 12 months after first-line chemoimmunotherapy to achieve CR;
   * Progression or relapse within 12 months after autologous hematopoietic stem cell transplantation;

     7. Life expectancy≥ 3 months 8. Clinical laboratory values meet screening visit criteria

   Exclusion Criteria:

   Subject eligible for this study must not meet any of the following criteria:
   1. Prior antitumor therapy with insufficient washout period ;
   2. Patients who received autologous CAR-T cell therapy (except CD19-targeted) or autologous gene therapy;
   3. Patients who received allogeneic hematopoietic stem cell transplantation or allogeneic therapy;

   5. Patients who are positive for any index of hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), or human immunodeficiency virus antibody (HIV- Ab).

   6. Known life-threatening allergies, hypersensitivity, or intolerance to LUCAR-G39P CAR-T cell or its excipients, including DMSO.

   7. Pregnant or lactating women;

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and type of TEAEs | Through study completion , an average of 2 years after LUCAR-G39P infusion (Day 1)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Pharmacokinetics in peripheral blood | ThTrough study completion , an average of 2 years after LUCAR-G39P infusion (Day 1)
  CAR positive T cells and CAR transgene levels in peripheral blood after LUCAR-G39P infusion
Pharmacokinetics in bone marrow | ThTrough study completion , an average of 2 years after LUCAR-G39P infusion (Day 1)
  CAR positive T cells and CAR transgene levels in bone marrow after LUCAR-G39P infusion.
The recommended Phase II dose (RP2D) for this cell therapy | Within 30 days after LUCAR-G39P infusion
  RP2D established through ATD+BOIN design and the DLTs occurring following CAR T-cell infusion

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, an average of 2 years after LUCAR-G39P infusion (Day 1)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via LUCAR-G39P cell infusion
Progression-free survival (PFS) | Through study completion, an average of 2 years after LUCAR-G39P infusion (Day 1)
  rogression Free Survival (PFS) is defined as the time from the date of first infusion of the LUCAR-G39P to the first documented disease progression (according to Lugano 2014) or death (due to any cause), whichever occurs first
Overall Survival (OS) | Through study completion, an average of 2 years after LUCAR-G39P infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LUCAR-G39P to death of the subject
Time to Response (TTR) | Through study completion, an average of 2 years after LUCAR-G39P infusion (Day 1)
  Time to Response (TTR) is defined as the time from the date of first infusion of LUCAR-G39P to the date of the first response evaluation of the subject who has met all criteria for CR or PR
Duration of Response (DoR) | Through study completion, an average of 2 years after LUCAR-G39P infusion (Day 1)
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (CR or PR) to the first documented relapse evidence of the responders.
Immunogenicity assessment of LUCAR-G39P cells | Through study completion, an average of 2 years after LUCAR-G39P infusion (Day 1)
  The incidence of Anti- LUCAR-G39P antibody in patients who received LUCAR-G39P cells infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, PhD,MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (3):
- China (3):
  - Department of Haematology, the First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjin, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Beijing Gobroad Hosptial, Beijing

IPD SHARING:
Plan to Share IPD: No